CLINICAL TRIAL: NCT03835260
Title: Pivot Breath Sensor Human Factors and Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Marler, MD (Industry)
Collaborators: UserWise, LLC (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Marler, MD, Senior Director, Clinical and Medical Affairs, Pivot Health Technologies Inc.
Organization: Pivot Health Technologies Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-404
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Smoking Cessation; Smoking, Tobacco
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pivot Breath Sensor (user group) (Other): Self-reported daily smokers of 2 or more cigarettes per day
  Interventions: Device: Pivot Breath Sensor

INTERVENTIONS:
Device: Pivot Breath Sensor — The Pivot Breath Sensor measures the level of carbon monoxide in exhaled breath and displays the carbon monoxide value to the user.

SUMMARY:
Prospective, observational open label, single center study enrolling up to 15 subjects to evaluate human factors and usability of the Pivot Breath Sensor.

DETAILED DESCRIPTION:
The objectives of this Human Factors/Usability study are to:

* Ensure that representative intended users are able to operate the Pivot Breath Sensor independently
* Validate appropriate mitigations of use related hazards identified in risk management documentation
* Uncover previously unforeseen use errors

This human factors and usability testing is conducted to demonstrate that the Pivot Breath Sensor can be used by the intended users without serious use errors or problems, for the intended uses and under the expected use conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* English speaking
* Owns and uses a smartphone
* Willing to sign the Informed Consent Form

Exclusion Criteria:

* Prior experience with a study sponsored by Carrot Inc
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Marler, MD, Principal Investigator — Pivot Health Technologies Inc.
Locations (1):
- Carrot Inc., Redwood City, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pivot Breath Sensor (User Group)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 15
Age, Customized [Count of Participants; unit: Participants]
  Age: Age 18-49 years | 13
  Age: Age 49-50 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 10
  Ethnicity: African American | 1
  Ethnicity: Middle Eastern | 2
  Ethnicity: Native American | 1
  Ethnicity: Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 15
Daily Smoking Frequency (cigarettes per day) [Count of Participants; unit: Participants]
  2-5 cpd | 2
  6-10 cpd | 4
  11-15 cpd | 4
  16+ cpd | 5

OUTCOME MEASURES:

1. Primary Outcome: Human Factors - User Performance in Use Scenarios Assessment With Observer Ratings
Description: User performance of participants in intended use scenarios will be assessed at a single visit. Participants will be observed if they can set up the device, use the device, and interpret results. Observer ratings include 'Successful' and 'Unsuccessful'. Specific attention will be given to assess if any harms can occur from observed use errors.
  'Successful' = user was able to complete the task safely and effectively. Unsuccessful' = user was unable unable to complete the task independently or did not complete the task safely and effectively.
  For each participant, the single visit includes the consent process, entry into the study, the study session, and conclusion of the study. The study session is completed on a single day requiring up to 60 minutes.
  Observations are made throughout the study session. Assessments for individual tasks will take approximately 1 minute and assessments will be made over the study session which can last up to 60 minutes.
Time Frame: Each study session was completed on a single day, for up to 60 minutes. Device set up was assessed at about 5 minutes in. Device use was assessed at about 10 minutes in. Interpretation of results was assessed at about 15 and 20 minutes in.
Measure: Count of Participants; unit: Participants
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 15
Participants
  Set up device - open packaging: Successful | 15
  Set up device - open packaging: Unsuccessful | 0
  Use device: Successful | 14
  Use device: Unsuccessful | 1
  Interpret results: Successful | 15
  Interpret results: Unsuccessful | 0

2. Primary Outcome: Human Factors - User Documentation Assessment With Observer Ratings
Description: Participant understanding of user documentation will be assessed at single visit. User documentation includes packaging information, quick start guide and user manual. Observer ratings include 'Successful' and 'Unsuccessful'.
  'Successful' = user was able to complete the task safely and effectively. Unsuccessful' = user was unable unable to complete the task independently or did not complete the task safely and effectively.
  For each participant, the single visit includes the consent process, entry into the study, the study session, and conclusion of the study. The study session is completed on a single day requiring up to 60 minutes.
  Observations are made throughout the study session. Assessments for individual tasks will take approximately 1 minute each. The User documentation assessment portion of the study session will last up to 30 minutes.
Time Frame: Each study session was completed on a single day, for up to 60 minutes. The user documentation assessment occurred at approximately 30 minutes into the study session.
Measure: Count of Participants; unit: Participants
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 15
Participants
  understanding of the packaging: Successful | 15
  understanding of the packaging: Unsuccessful | 0
  understanding of the quick start guide: Successful | 14
  understanding of the quick start guide: Unsuccessful | 1
  understanding of the user manual: Successful | 15
  understanding of the user manual: Unsuccessful | 0

3. Primary Outcome: Human Factors - Subjective Feedback Questionnaire
Description: Subjective feedback focusing on any concerns on using device will be assessed at single visit. Participants will answer with a Yes or No to the questions.
  For each participant, the single visit includes the consent process, entry into the study, the study session, and conclusion of the study. The study session is completed on a single day requiring up to 60 minutes.
  Subjective feedback focusing on any concerns prior to the conclusion of the study session. Subjective feedback questions will take approximately 1-3 minutes each. The Subjective feedback portion of the study session will last up to 5 to 15 minutes.
Time Frame: Each study session was completed on a single day, for up to 60 minutes. The subjective feedback questionnaire was administered at approximately 40 minutes into the study session.
Measure: Count of Participants; unit: Participants
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 15
Participants
  Dd you experience any moments of hesitation while using the product?: yes | 10
  Dd you experience any moments of hesitation while using the product?: no | 5
  Do you have any safety concerns regarding this product or its labeling?: yes | 3
  Do you have any safety concerns regarding this product or its labeling?: no | 12

4. Primary Outcome: Human Factors - Participant Feedback Using Rating Scale
Description: Participant will be asked to provide ratings on the following:
  * How would you rate the ease or difficulty using the device?
  * How clear or unclear was the Quick Start Guide?
  * How clear or unclear was the Packaging?
  * How clear or unclear was the User Manual?
  * How easy or difficult was it to understand and interpret the test results?
  The participant will use the following rating scale (higher score = better outcome):
  5 - Very Easy 4 - Easy 3 - Neither Easy nor Difficult 2 - Difficult
  1 - Very difficult
  For each participant, the single visit includes the consent process, entry into the study, the study session, and conclusion of the study. The study session is completed on a single day requiring up to 60 minutes.
  Participant will provide the ratings prior to the conclusion of the study session. Participant assessment with questionnaire rating scales will take approximately 1-2 minutes each.
Time Frame: Each study session was completed on a single day, for up to 60 minutes. Participant feedback using a rating scale was provided at approximately 50 minutes into the study session.
Measure: Count of Participants; unit: Participants
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 15
Participants
  How would you rate the ease or difficulty of using the device?: very easy/very clear | 5
  How would you rate the ease or difficulty of using the device?: easy/clear | 8
  How would you rate the ease or difficulty of using the device?: neither easy/clear nor difficult/unclear | 2
  How would you rate the ease or difficulty of using the device?: difficult/unclear | 0
  How would you rate the ease or difficulty of using the device?: very difficult/very unclear | 0
  How clear or unclear was the Quick Start Guide?: very easy/very clear | 8
  How clear or unclear was the Quick Start Guide?: easy/clear | 6
  How clear or unclear was the Quick Start Guide?: neither easy/clear nor difficult/unclear | 1
  How clear or unclear was the Quick Start Guide?: difficult/unclear | 0
  How clear or unclear was the Quick Start Guide?: very difficult/very unclear | 0
  How clear or unclear was the packaging?: very easy/very clear | 9
  How clear or unclear was the packaging?: easy/clear | 5
  How clear or unclear was the packaging?: neither easy/clear nor difficult/unclear | 1
  How clear or unclear was the packaging?: difficult/unclear | 0
  How clear or unclear was the packaging?: very difficult/very unclear | 0
  How clear or unclear was the User Manual on the iPad?: very easy/very clear | 11
  How clear or unclear was the User Manual on the iPad?: easy/clear | 4
  How clear or unclear was the User Manual on the iPad?: neither easy/clear nor difficult/unclear | 0
  How clear or unclear was the User Manual on the iPad?: difficult/unclear | 0
  How clear or unclear was the User Manual on the iPad?: very difficult/very unclear | 0
  How easy or difficult was it to understand and interpret the test results?: very easy/very clear | 5
  How easy or difficult was it to understand and interpret the test results?: easy/clear | 8
  How easy or difficult was it to understand and interpret the test results?: neither easy/clear nor difficult/unclear | 2
  How easy or difficult was it to understand and interpret the test results?: difficult/unclear | 0
  How easy or difficult was it to understand and interpret the test results?: very difficult/very unclear | 0

ADVERSE EVENTS:
Time Frame: Adverse events were observed for throughout the entirety of each participant's study session, up to 60 minutes during a session on one day.
Arm/Group | Pivot Breath Sensor (User Group)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT03835260/Prot_SAP_001.pdf